CLINICAL TRIAL: NCT03805737
Title: Indoor Daylight Photo Dynamic Therapy (PDT) for Actinic Keratosis
Brief Title: Indoor Daylight Photo Dynamic Therapy for Actinic Keratosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Norris Cotton Cancer Center (Other)
Responsible Party: Principal Investigator, Michael S. Chapman, Staff Physican, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D19030
Record Dates: First submitted 2019-01-14; First posted 2019-01-16 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — Sunlight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Indoor Daylight PDT Therapy (Experimental): Ameluz will be applied to skin. This will be followed by a 30-minute incubation period. Subsequently, you will be exposed to natural sunlight through a window for 2 hours. Post-treatment assessments will be performed and you will be given instruction on appropriate sun protection methods.
  Interventions: Other: Amulez and sunlight
- FDA Approved Standard Light Therapy Treatment (Active Comparator): Ameluz will be applied to skin. This will be followed by a 30-minute incubation period. Subsequently, you will receive Red Light Treatment for 10 minutes. Post-treatment assessments will be performed and you will be given instruction on appropriate sun protection methods.
  Interventions: Other: Amulez and red light treatment

INTERVENTIONS:
Other: Amulez and sunlight — Amulez and sun exposure for 2 hours
  Arms: Indoor Daylight PDT Therapy
Other: Amulez and red light treatment — Amulez and red light treatment for 10 minutes
  Arms: FDA Approved Standard Light Therapy Treatment

SUMMARY:
The purpose of this study is to understand better if indoor daylight Photo Dynamic Therapy (PDT) can provide effective lesion clearing versus conventional red lamp light therapy.

DETAILED DESCRIPTION:
Subjects who enroll into this research study, their participation in this study will last up to 6 months. They will be asked to return to the clinic 3-4 times.

Subjects will be randomized into one of two study arms:

Arm 1 - Indoor Daylight PDT Therapy Arm 2 - FDA Approved Standard Light Therapy Treatment

ELIGIBILITY:
Inclusion Criteria:

* All patients with actinic keratosis appearing at the Dermatology Clinic for PDT treatment.
* Age ≥ 18 years older.

Exclusion Criteria:

* Pregnant women or women who are breast-feeding.
* Any patients with a condition that makes them not suitable for clinical PDT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-10-06 (Actual); Study Completion 2021-10-06 (Actual)

PRIMARY OUTCOMES:
Changes or clearing of the lesions | Baseline, immediately post-procedure (2 hours) and one and 6 months
  The primary aim of this study is to study if indoor daylight PDT can be as effective as regular lamp light PDT. This study can be confounded by the amount of PpIX produced in the lesions as well as the clearing of lesions at one month and six months.
Change in the amount of PpIX in the lesion | Baseline and immediately post procedure
  Secondary diagnostic study to determine if low-cost cellphone-based skin dosimetry in PDT can facilitate objective measurement of drug levels.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Shane Chapman, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhao B, He YY. Recent advances in the prevention and treatment of skin cancer using photodynamic therapy. Expert Rev Anticancer Ther. 2010 Nov;10(11):1797-809. doi: 10.1586/era.10.154. PMID 21080805
- [Background] Wiegell SR, Wulf HC, Szeimies RM, Basset-Seguin N, Bissonnette R, Gerritsen MJ, Gilaberte Y, Calzavara-Pinton P, Morton CA, Sidoroff A, Braathen LR. Daylight photodynamic therapy for actinic keratosis: an international consensus: International Society for Photodynamic Therapy in Dermatology. J Eur Acad Dermatol Venereol. 2012 Jun;26(6):673-9. doi: 10.1111/j.1468-3083.2011.04386.x. Epub 2011 Dec 23. PMID 22211665
- [Background] Griffin LL, Lear JT. Photodynamic Therapy and Non-Melanoma Skin Cancer. Cancers (Basel). 2016 Oct 22;8(10):98. doi: 10.3390/cancers8100098. PMID 27782094
- [Background] Zhao SG, Chen XF, Wang LG, Yang G, Han DY, Teng L, Yang MC, Wang DY, Shi C, Liu YH, Zheng BJ, Shi CB, Gao X, Rainov NG. Increased expression of ABCB6 enhances protoporphyrin IX accumulation and photodynamic effect in human glioma. Ann Surg Oncol. 2013 Dec;20(13):4379-88. doi: 10.1245/s10434-011-2201-6. Epub 2012 Jun 12. PMID 22688660
- [Background] Tyrrell JS, Morton C, Campbell SM, Curnow A. Comparison of protoporphyrin IX accumulation and destruction during methylaminolevulinate photodynamic therapy of skin tumours located at acral and nonacral sites. Br J Dermatol. 2011 Jun;164(6):1362-8. doi: 10.1111/j.1365-2133.2011.10265.x. Epub 2011 May 13. PMID 21564050
- [Background] Nissen CV, Philipsen PA, Wulf HC. Protoporphyrin IX formation after topical application of methyl aminolaevulinate and BF-200 aminolaevulinic acid declines with age. Br J Dermatol. 2015 Sep;173(3):760-6. doi: 10.1111/bjd.13923. Epub 2015 Aug 20. PMID 25997508
- [Background] Kanick SC, Davis SC, Zhao Y, Hasan T, Maytin EV, Pogue BW, Chapman MS. Dual-channel red/blue fluorescence dosimetry with broadband reflectance spectroscopic correction measures protoporphyrin IX production during photodynamic therapy of actinic keratosis. J Biomed Opt. 2014;19(7):75002. doi: 10.1117/1.JBO.19.7.075002. PMID 24996661
- [Background] Kanick SC, Davis SC, Zhao Y, Sheehan KL, Hasan T, Maytin EV, Pogue BW, Chapman MS. Pre-treatment protoporphyrin IX concentration in actinic keratosis lesions may be a predictive biomarker of response to aminolevulinic-acid based photodynamic therapy. Photodiagnosis Photodyn Ther. 2015 Dec;12(4):561-6. doi: 10.1016/j.pdpdt.2015.10.006. Epub 2015 Oct 22. PMID 26480810
- [Background] Pogue BW, Burke G. Fiber-optic bundle design for quantitative fluorescence measurement from tissue. Appl Opt. 1998 Nov 1;37(31):7429-36. doi: 10.1364/ao.37.007429. PMID 18301577
- [Derived] Ruiz AJ, LaRochelle EPM, Fahrner MP, Emond JA, Samkoe KS, Pogue BW, Chapman MS. Equivalent efficacy of indoor daylight and lamp-based 5-aminolevulinic acid photodynamic therapy for treatment of actinic keratosis. Skin Health Dis. 2023 Mar 31;3(4):e226. doi: 10.1002/ski2.226. eCollection 2023 Aug. PMID 37538332